CLINICAL TRIAL: NCT00347009
Title: An Open Label Study of Adefovir Dipivoxil for the Treatment of Patients With Chronic Hepatitis B Related Advanced Fibrosis or Cirrhosis.
Brief Title: Adefovir Dipivoxil For The Treatment Of Patients With Chronic Hepatitis B Related Advanced Fibrosis Or Cirrhosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADF104070
Record Dates: First submitted 2006-06-30; First posted 2006-07-04 (Estimated); Results first posted 2010-10-15 (Estimated); Last update posted 2012-06-04 (Estimated); Status verified 2011-03

CONDITIONS: Hepatitis B, Chronic; Cirrhosis; Fibrosis; Chronic Hepatitis B
Keywords: Cirrhosis; Advanced Fibrosis; Chronic Hepatitis B; Adefovir Dipivoxil
MeSH Terms: conditions — Hepatitis B, Chronic; Fibrosis | interventions — adefovir dipivoxil

ARMS (1):
- Adefovir Dipivoxil (Other): 10mg once daily in patients with CHB related advanced fibrosis/cirrhosis.
  Interventions: Drug: adefovir dipivoxil

INTERVENTIONS:
Drug: adefovir dipivoxil — 10mg once daily

SUMMARY:
This 36-month open-label study of adefovir dipivoxil investigates the clinical benefits of the therapy in chronic hepatitis B patients with advanced fibrosis or cirrhosis confirmed with biopsy. Primary endpoint is histological improvement defined as a decrease of Ishak Fibrosis Score by one point or more from baseline at Month 36 of adefovir dipivoxil treatment. Approximately 150 patients will be recruited in study centres in the Asia Pacific area. The patients are offered 36 months of open label adefovir dipivoxil treatment, with assessments every three months, after which there is a 6-month post study treatment follow-up prior to study completion. After the 36 months of study treatment, it is likely that the patient will benefit from continued treatment with adefovir dipivoxil. If this is the case in the investigators clinical judgement, the investigator should ensure that a routine prescription is available in a timely manner, and that no unnecessary interruption in treatment occurs.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients ≥ 18 years of age
* A female is eligible to enter and participate in this study if she is of: a) non-childbearing potential (ie. Physiologically incapable of becoming pregnant, including any female who is pre-menarchal or post-menopausal); b) child-bearing potential with a negative serum pregnancy test at screen, and agrees to one of the following: -complete abstinence from intercourse from 2 weeks prior to administration of the study drug, throughout the study, and for a time interval after completion or premature discontinuation from the study to account for elimination of the investigational drug, (a minimum of 5 half-lives or longer if the pharmacodynamic profile of the investigational drug warrants a longer time period); or, -Female sterilization; or -Sterilization of male partner; or -Implants of levonorgestrel; or, -Injectable progestogen; or -Oral contraceptive (combined or progestogen only); or, -Any intrauterine device (IUD) with published data showing that the lowest expected failure rate is less that 1% per year (not all IUDs meet this criterion); or, -Any other methods with published data showing that the lowest expected failure rate for that method is less than 1% per year; or, -Barrier method only if used in combination with any of the above acceptable methods.
* Documented chronic hepatitis B infection determined by presence of serum HBsAg for at least 6 months (positive once at least 6 months before screening and at time of screening visit.)
* Positive HBV DNA plasma assay with screening value ≥ 1 x 10^5 copies /mL. (Roche COBAS AMPLICOR TM HBV Monitor Test, LLOD <300 copies/mL )
* Adequate renal function defined as serum creatinine ≤1.5 mg/dL (≤130 µmol/L).
* Willing and able to undergo two liver biopsies (prior to dosing, and after 36 months of therapy). The study baseline liver biopsy can be the most recent liver biopsy taken within 6 months of enrollment, as long as the biopsy was taken 6 months or more after the completion of any interferon or 3 months or more after completion of any antiviral treatment (eg. famciclovir, lamivudine etc.), and the patient has not had interferon therapy or any antiviral therapy between the biopsy and screening.
* Liver biopsy showing advance fibrosis/cirrhosis (Ishak fibrosis score ≥4). The slides must be available for review by an independent histopathologist.
* Availability and willingness of the subject to provide written informed consent per ICH/GCP and local Guidelines.

Exclusion Criteria:

1. ALT >10XULN at screening
2. Child-Pugh Score ≥ 7
3. History of acute exacerbation leading to transient decompensation
4. Co-infections with HIV, HCV or HDV. Note: Patients who are anti-HCV seropositive and in whom HCV RNA is undetectable are considered to be HCV seropositive and will not be eligible for enrollment.
5. Any of the following laboratory parameter within 4 weeks prior to study entry: -Haemoglobin <8.0 g/dL, -Absolute neutrophil count (ANC) < 1.5 x 10^9/L, -Platelet count ≤50 x 10^9/L, -Pancreatic amylase and/or lipase >2 x ULN

   * Screening alpha-fetoprotein (AFP) value >50 ng/mL
   * Clinical, ultrasonographic or radiologic evidence of hepatic mass suggestive of hepatocellular carcinoma.
   * Significant concurrent medical and/or psychiatric conditions other than hepatitis B that in the opinion of the investigators might interfere with patient's treatment, assessment or compliance according to study requirement, such as malignancy, congestive heart failure, renal failure, chronic pancreatitis, diabetes mellitus with poor control and alcoholism.
   * Any of the following medications with 2 months prior to study entry (or the expectation that subject will receive these during the course of the study): -Nephrotoxic medication (eg aminoglycosides, amphotericin B, vancomycin, cidofovir, foscarnet, cisplatin, pentamidine) or competitors or renal excretion (eg probenecid, sulfinpyrazone), -Hepatotoxic medication (eg anabolic steroids,ketoconazole, itraconazole, isoniazid, rifampin, rifabutin).
   * Treatment with immunosuppressive/immunomodulatory agents (including interferon and corticosteroids) within 6 months prior to study entry.
   * Presence of other causes of liver disease (ie. hemochromatosis, Wilson's disease, alcoholic liver disease, non-alcoholic steatohepatitis, autoimmune hepatitis, alpha-1 antitrypsin deficiency).
   * A history of liver transplantation /planned for liver transplantation.
   * Pregnancy (or lactation) or , in subjects capable of bearing children, inability/unwillingness to practice adequate contraception.
   * Females of child-bearing potential (post-puberty) willing or unable to have pregnancy testing at any study visit.
   * History of hypersensitivity to nucleoside and/or nucleotide analogues.
   * Concurrent participation in another clinical trial in which the subject is or will be exposed to another investigational or a non-investigational drug or device within 30 days of the screening visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2005-05; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (9):
- GSK Investigational Site, Pokfulam, Hong Kong
- GSK Investigational Site, Singapore, Singapore
- South Korea (4):
  - GSK Investigational Site, Daegu
  - GSK Investigational Site, Pusan
  - GSK Investigational Site, Seoul
  - GSK Investigational Site, Sungnam-City
- Taiwan (2):
  - GSK Investigational Site, Kaohsiung City
  - GSK Investigational Site, Taipei
- GSK Investigational Site, Ho Chi Minh City, Vietnam

RESULTS

PARTICIPANT FLOW:
Groups:
- Adefovir Dipivoxil 10 Milligrams (mg): Adefovir Dipivoxil 10 mg, once daily
Period: Overall Study
Arm/Group | Adefovir Dipivoxil 10 Milligrams (mg)
Started | 155
Completed | 128
Not Completed | 27
Not completed — Death | 1
Not completed — Adverse Event | 6
Not completed — Withdrawal by Subject | 3
Not completed — Physician Decision | 5
Not completed — Lost to Follow-up | 4
Not completed — Protocol Violation | 2
Not completed — Adverse Laboratory Experience | 1
Not completed — Insufficient Viral Suppression | 3
Not completed — Increased ALT/HBV DNA | 1
Not completed — Serious Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Adefovir Dipivoxil 10 Milligrams (mg)
Number analyzed (Participants) | 155
Age Continuous [Mean (Standard Deviation); unit: Years] | 47.7 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39
  Male | 116
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 155
  Other | 0
Time since Diagnosis of Chronic Hepatitis B [Mean (Standard Deviation); unit: years] — Diagnosis of chronic hepatitis B is defined by the presence of serum hepatitis B surface antigen (HBsAg) for at least 6 months (once at least 6 months before screening and at time of screening visit).
  years | 11.29 (8.40)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Histologic Improvement at Month 36 (Intent-to-Treat Population)
Description: The Ishak fibrosis score is a scoring system (ranging from 0 to 6) that measures the degree of fibrosis (scarring) of the liver, which is caused by chronic necroinflammation (an inflammatory process in the liver including or leading to death of liver cells). A score of 0 represents no fibrosis, and a score of 6 represents established cirrhosis. Participants were classified as improved if the Ishak fibrosis score at Month 36 was 1 or more points less from the Screening score.
Time Frame: Screening and Month 36
Population: Intent-to-Treat (ITT) Population: all participants who received at least one dose of study medication, regardless of whether the participants completed the planned duration of the study
Measure: Number; unit: participants
Arm/Group | Adefovir Dipivoxil 10 Milligrams (mg)
Number analyzed (Participants) | 155
participants | 52

2. Secondary Outcome: Number of Participants With a Reduction From Baseline in the Child-Pugh Score by 2 Points or More at Months 12, 24, and 36
Description: The Child-Pugh score (modified version for scoring prothrombin time against reference range) was used in the study to assess the prognosis of chronic liver disease, mainly cirrhosis. The score employs five clinical measures of liver disease: encephalopathy, ascites, albumin, prothrombin time, and bilirubin. Each measure is scored on a scale of 1-3, with 1 being normal and 3 indicating most severe derangement. The total score for the Child-Pugh assessment was calculated as the sum of the 5 contributing scores, with a score range of 5 (best prognosis) to 15 (worst prognosis).
Time Frame: Baseline and Months 12, 24, and 36
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Adefovir Dipivoxil 10 Milligrams (mg)
Number analyzed (Participants) | 155
participants
  Month 12 | 0
  Month 24 | 2
  Month 36 | 1

3. Secondary Outcome: Number of Participants With a Reduction From Screening of at Least 2 Points in the Knodell Necroinflammation Score at Month 36
Description: The Knodell scoring system, also called the Histologic Activity Index (HAI), classifies liver biopsy specimens according to scores into 4 categories of histologic features: (I) periportal and/or bridging necrosis (scores from 0 to 10); (II) intralobular degeneration and focal necrosis (scores from 0 to 4); (III) portal inflammation (scores from 0 to 4); (IV) fibrosis (scores from 0 to 4). The Knodell necroinflammation score is the sum of scores from Parts I-III, hence a range of 0 to 18, and measures the degree of acute necroinflammatory activity in the liver.
Time Frame: Screening and Month 36
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Adefovir Dipivoxil 10 Milligrams (mg)
Number analyzed (Participants) | 155
participants | 64

4. Secondary Outcome: Change From Baseline in Serum Hepatitis B Virus (HBV) Deoxyribonucleic Acid (DNA) Level at Months 12, 24, and 36
Description: The levels of HBV DNA in serum were measured using the Amplicor Cobas assay by Roche Diagnostics (detection limit 300 copies/milliliter [ml]). Changes from baseline in the serum HBV DNA level at Months 12, 24 and 36 were calculated as Month 12 minus baseline, Month 24 minus baseline, and Month 36 minus baseline respectively. Change is reported in log10 units.
Time Frame: Baseline and Months 12, 24, and 36
Population: ITT Population
Measure: Mean (Standard Deviation); unit: log10 copies/ml
Arm/Group | Adefovir Dipivoxil 10 Milligrams (mg)
Number analyzed (Participants) | 155
log10 copies/ml
  Month 12 | -4.557 (1.639)
  Month 24 | -4.536 (2.115)
  Month 36 | -4.454 (2.436)

5. Secondary Outcome: Number of Participants Achieving Virological Response (HBV DNA Level <= 10^3 Copies/ml) at Months 12, 24, and 36
Description: Virological response was defined as an HBV DNA level <= 10^3 copies/ml.
Time Frame: Months 12, 24, and 36
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Adefovir Dipivoxil 10 Milligrams (mg)
Number analyzed (Participants) | 155
participants
  Month 12 | 91
  Month 24 | 99
  Month 36 | 102

6. Secondary Outcome: Number of Participants Achieving Virological Response (HBV DNA Level <= 10^4 Copies/ml) at Months 12, 24, and 36
Description: Virological response was defined as an HBV DNA level <= 10^4 copies/ml.
Time Frame: Months 12, 24, and 36
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Adefovir Dipivoxil 10 Milligrams (mg)
Number analyzed (Participants) | 155
participants
  Month 12 | 110
  Month 24 | 114
  Month 36 | 109

7. Secondary Outcome: Number of Participants With Undetectable HBV DNA at Months 12, 24, and 36
Description: Undetectable HBV DNA was defined as an HBV DNA level below the lower limit of detection (LLOD) of 300 copies/ml.
Time Frame: Months 12, 24, and 36
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Adefovir Dipivoxil 10 Milligrams (mg)
Number analyzed (Participants) | 155
participants
  Month 12 | 83
  Month 24 | 95
  Month 36 | 90

8. Secondary Outcome: Number of Participants With Virological Breakthrough at Months 12, 24, and 36
Description: Virological breakthrough was defined as an increase in serum HBV DNA levels by more than 1 log10 copies/ml from treatment nadir, i.e., the lowest HBV DNA value during the study.
Time Frame: Months 12, 24, and 36
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Adefovir Dipivoxil 10 Milligrams (mg)
Number analyzed (Participants) | 155
participants
  Month 12 | 3
  Month 24 | 16
  Month 36 | 21

9. Secondary Outcome: Number of Participants With Alanine Aminotransferase (ALT) Normalization at Months 12, 24, and 36
Description: ALT levels were measured as part of the liver function tests. Participants with ALT normalization at each visit were defined as those with a value below the upper limit of the normal (ULN) range for ALT provided by that site at the respective visit.
Time Frame: Months 12, 24, and 36
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Adefovir Dipivoxil 10 Milligrams (mg)
Number analyzed (Participants) | 155
participants
  Month 12 | 87
  Month 24 | 91
  Month 36 | 91

10. Secondary Outcome: Number of Participants Who Were Hepatitis B Envelope Antigen (HBeAg) Positive at Baseline and Developed Undetectable Levels of HBeAg at Months 12, 24, and 36
Description: HBeAg positive was defined as the presence of a detectable level of HBeAg.
Time Frame: Baseline and Months 12, 24, and 36
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Adefovir Dipivoxil 10 Milligrams (mg)
Number analyzed (Participants) | 155
participants
  Month 12 | 17
  Month 24 | 27
  Month 36 | 28

11. Secondary Outcome: Number of Participants Who Were HBeAg Positive at Baseline, With HBeAg Seroconversion at Months 12, 24, and 36
Description: HBeAg seroconversion was defined as a decrease in HBeAg to undetectable levels and a gain of detectable levels of Hepatitis B envelope antibody (HBeAb).
Time Frame: Baseline and Months 12, 24, and 36
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Adefovir Dipivoxil 10 Milligrams (mg)
Number analyzed (Participants) | 155
participants
  Month 12 | 10
  Month 24 | 18
  Month 36 | 15

12. Secondary Outcome: Number of Participants Who Were Hepatitis B Surface Antigen (HBsAg) Positive at Baseline and Developed Undetectable Levels of HBsAg at Months 12, 24, and 36
Description: HBsAg positive was defined as the presence of a detectable level of HBsAg.
Time Frame: Baseline and Months 12, 24, and 36
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Adefovir Dipivoxil 10 Milligrams (mg)
Number analyzed (Participants) | 155
participants
  Month 12 | 0
  Month 24 | 0
  Month 36 | 0

13. Secondary Outcome: Number of Participants Who Were HBsAg Positive at Baseline, With HBsAg Seroconversion at Months 12, 24, and 36
Description: HBsAg seroconversion was defined as a decrease in HBsAg to undetectable levels and a gain of detectable levels of Hepatitis B surface antibody (HBsAb).
Time Frame: Baseline and Months 12, 24, and 36
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Adefovir Dipivoxil 10 Milligrams (mg)
Number analyzed (Participants) | 155
participants
  Month 12 | 0
  Month 24 | 0
  Month 36 | 0

14. Primary Outcome: Number of Participants With Histologic Improvement at Month 36 (Per Protocol Population)
Description: as for outcome 1
Time Frame: Screening and Month 36
Population: Per Protocol (PP) Population: all participants in the ITT Population with interpretable liver biopsies at baseline and at the 36-month follow-up visit and without major violations of the protocol
Measure: Number; unit: participants
Arm/Group | Adefovir Dipivoxil 10 Milligrams (mg)
Number analyzed (Participants) | 114
participants | 52

ADVERSE EVENTS:
Time Frame: Screening to Month 42
Description: Adverse events (AEs) were reported spontaneously by the participant or determined by the investigator through questioning the participant in a general way; the severity, outcome and cause of each reported AE were assessed and recorded.
Arm/Group | Adefovir Dipivoxil 10 Milligrams (mg)
Serious Adverse Events (participants affected / at risk) | 20/155
Other Adverse Events (participants affected / at risk) | 99/155
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adefovir Dipivoxil 10 Milligrams (mg) (N=155)
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7
Hepatic neoplasm malignant recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Cerebellar tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Duodenal ulcer (Gastrointestinal disorders) | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 1
Oesophageal obstruction (Gastrointestinal disorders) | 1
Drug exposure during pregnancy (Injury, poisoning and procedural complications) | 1
Excoriation (Injury, poisoning and procedural complications) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
Ribs fracture (Injury, poisoning and procedural complications) | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1
Acute sinusitis (Infections and infestations) | 1
Appendicitis (Infections and infestations) | 1
Hepatitis B (Infections and infestations) | 1
Periorbital cellulitis (Infections and infestations) | 1
Pneumonia bacterial (Infections and infestations) | 1
Bile duct stone (Hepatobiliary disorders) | 1
Cholangitis (Hepatobiliary disorders) | 1
Jaundice cholestatic (Hepatobiliary disorders) | 1
Hepatic encephalopathy (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 1
Depression (Psychiatric disorders) | 1
Suicide attempt (Psychiatric disorders) | 1
Diabetic nephropathy (Renal and urinary disorders) | 1
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Adefovir Dipivoxil 10 Milligrams (mg) (N=155)
Abdominal pain upper (Gastrointestinal disorders) | 15
Diarrhoea (Gastrointestinal disorders) | 11
Abdominal distension (Gastrointestinal disorders) | 10
Gastritis (Gastrointestinal disorders) | 9
Upper respiratory tract infection (Infections and infestations) | 40
Back pain (Musculoskeletal and connective tissue disorders) | 12
Cough (Respiratory, thoracic and mediastinal disorders) | 16
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 9
Fatigue (General disorders) | 13
Alanine aminotransferase increased (Investigations) | 26
Aspartate aminotransferase increased (Investigations) | 23
Hepatitis B DNA increased (Investigations) | 9
Alpha 1 fetoprotein increased (Investigations) | 8
Pruritus (Skin and subcutaneous tissue disorders) | 10
Headache (Nervous system disorders) | 8
Insomnia (Psychiatric disorders) | 8
Hypertension (Vascular disorders) | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.